CLINICAL TRIAL: NCT03855098
Title: Identification of New Dietary Biomarkers Using a Cross-over Feeding Study Among 25 Individuals in University College Dublin
Brief Title: Biomarkers of Food Intake Using a Cross-over Feeding Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Dublin (Other)
Responsible Party: Principal Investigator, Lorraine Brennan, Principle Investigator, University College Dublin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UCD_123_2019
Record Dates: First submitted 2019-02-19; First posted 2019-02-26 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-05

CONDITIONS: Diet Habit
Keywords: Metabolomics; dietary biomarkers; personalized nutrition
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Intervention Model Description: Each participant is asked to eat a test food (mixed vegetables (spinach and lettuce), green beans and mixed berries (strawberries and blueberries). They are asked for urine samples for up to 6 hours after eating each food. They are also asked for a urine sample one day after eating the foods. The samples are then analysed for dietary biomarkers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fruit and Vegetable biomarkers (Other): Each participant will consume the test foods over different weeks
  Interventions: Other: Biomarkers of Fruit and Vegetable Intake

INTERVENTIONS:
Other: Biomarkers of Fruit and Vegetable Intake — Cross-over study where participants will visit the Human Intervention Centre (in UCD) on 3 occasions (3 study days) with a minimum one week between each visit. The order of consumption of the test foods will be randomized. The test foods are mixed vegetables (spinach and lettuce), green beans and mixed berried (strawberries and blueberries). The following definition of portion sizes will be used; green beans (120g), lettuce (20g), spinach (90g), strawberries (96g) and blueberries (75g).
  For each study day, the participants will arrive fasting and provide a urine sample (0h sample). For 24h prior to the study day participants will avoid the test foods. Participants will consume the food and urine samples will be taken at 2, 4, 6 and 24 h post consumption.

SUMMARY:
Assessment of dietary intake is key for understanding the links between diet and health. Here, researchers will study molecules in urine samples to give them an insight into what people have eaten. These new molecules are called dietary biomarkers. This study will help to identify new molecules that can act as biomarkers of commonly consumed foods. These can then be used in the assessment of diet, identification of diet-related diseases and used how to explain how a dietary intervention (programme) will work, thereby adding to scientific knowledge.

DETAILED DESCRIPTION:
For biomarker discovery a cross-over study where participants will visit the Human Intervention Centre (in UCD) on 3 occasions (3 study days) with a minimum one week between each visit. The order of consumption of the test foods will be randomized. The test foods are mixed vegetables (spinach and lettuce), green beans and mixed berried (strawberries and blueberries). For each study day, the participants will arrive fasting and provide a urine sample (0h sample). For 24h prior to the study day participants will avoid the test foods. Participants will consume the food and urine samples will be taken at 2, 4, 6 and 24 h post consumption . Standard portions of the test food will be eaten on each occasion. Between the visits, participants will consume their habitual diet.

The samples will be analysed using the metabolomics platforms LC-MS and NMR spectroscopy. Both NMR and LC-MS data generated will undergo statistical analysis such as principal component analysis (PCA) and supervised analysis such as partial least squares-discriminant analysis (PLS-DA). Validation of such models will be performed using permutation testing.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults aged 18-50 years old
2. BMI<30.

Exclusion Criteria:

1. Smokers
2. Diagnosed health condition (chronic or infectious disease)
3. Taking medication (oral contraceptive pill is allowed)
4. Pregnant, lactating
5. Allergies/intolerances to any of specified test foods

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-20 (Actual)

PRIMARY OUTCOMES:
Urinary biomarker changes following consumption of specific foods will be measured using metabolomic approaches in post consumption samples. | 2, 4 and 6 hours post consumption of the test food. Urine samples are taken postprandially to determine how the biomarkers behave post consumption, which is standard practice in dietary biomaker identification studies.
  A number of biomarkers will be identified for the test foods. These biomarkers will be measured using LC/MS and NMR spectroscopy and will be reported in relative units. An untargeted approach will be applied to measure the biomarkers, of which hundreds will be measured. These biomarkers will be from different classes of compounds such as amino acids, fatty acids, lipids and carbohydrates for example.
  Note: A list of biomarkers has not been added as the investigators are using an untargeted metabolomics approach, which will be used to identify biomarkers from different compound classes.

CONTACTS AND LOCATIONS:
Overall Officials: Lorraine Brennan, PhD, Principal Investigator — University College Dublin
Locations (1):
- University College Dublin, Dublin, Dublin 4, Ireland

IPD SHARING:
Plan to Share IPD: No